CLINICAL TRIAL: NCT00388726
Title: The "EMBRACE" Trial: Eisai Metastatic Breast Cancer Study Assessing Physician's Choice Versus E7389. A Phase III Open-Label, Randomized, Parallel, Two-arm, Multi-center Study of E7389 Versus "Treatment of Physician's Choice" in Patients With Locally Recurrent, Metastatic Breast Cancer, Previously Treated With At Least Two and a Maximum of Five Prior Chemotherapy Regimens, Including an Anthracycline and a Taxane
Brief Title: E7389 Versus Treatment of Physician's Choice in Patients With Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Eisai Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7389-G000-305; 2006-001949-34 (EudraCT Number)
Record Dates: First submitted 2006-10-13; First posted 2006-10-17 (Estimated); Results first posted 2012-01-30 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2014-07

CONDITIONS: Breast Cancer
Keywords: Locally recurrent breast cancer; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: E7389
- 2 (Active Comparator)
  Interventions: Drug: Physician's Choice

INTERVENTIONS:
Drug: E7389 — 1.4 mg/m^2 intravenous (IV) infusion given over 2-5 minutes on Days 1 and 8 every 21 days.
  Arms: 1
Drug: Physician's Choice — Treatment of the Physician's Choice defined as any single agent chemotherapy, hormonal treatment or biological therapy approved for the treatment of cancer; or palliative treatment or radiotherapy, administered according to local practice, if applicable.
  Arms: 2

SUMMARY:
The purpose of this study is to compare Overall Survival (OS), Progression Free Survival (PFS), objective tumor response rate, duration of response, and safety in patients treated with E7389 versus the Treatment of Physician's Choice (TPC) in patients with locally recurrent or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with histologically or cytologically confirmed carcinoma of the breast.

   Every effort should be made to make paraffin embedded tissue or slides from the diagnostic biopsy or surgical specimen available for confirmation of diagnosis.
2. Patients with locally recurrent or metastatic disease who have received at least two (and not more than five) prior chemotherapeutic regimens for breast cancer, at least two of which were administered for treatment of locally recurrent and/or metastatic disease.

   Prior therapy must be documented by the following criteria prior to entry onto study:
   * Regimens must have included an anthracycline (e.g., doxorubicin, epirubicin) and a taxane (e.g., paclitaxel, docetaxel) in any combination or order. Treatment with any of these agents is not required if they are contraindicated for a certain patient.
   * One or two of these regimens may have been administered as adjuvant and/or neoadjuvant therapy, but at least 2 must have been given for relapsed or metastatic disease.
   * Patients must have proved refractory to the most recent chemotherapy, documented by progression on or within six (6) months of therapy.
   * Patients with Human Epidermal Growth Factor 2 (HER2/neu) positive tumors may additionally have been treated with trastuzumab.
   * Patients may have additionally been treated with anti-hormonal therapy.
3. Resolution of all chemotherapy or radiation-related toxicities to Grade 1 severity or lower, except for stable sensory neuropathy <= Grade 2 and alopecia.
4. Age >= 18 years.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2.
6. Life expectancy of >= 3 months.
7. Adequate renal function as evidenced by serum creatinine <= 2.0 mg/dL or calculated creatinine clearance >= 40 mL/min per the Cockcroft and Gault formula.
8. Adequate bone marrow function as evidenced by absolute neutrophil count (ANC) >= 1.5 x 10^9/L, hemoglobin >= 10.0 g/dL (a hemoglobin <10.0 g/dL is acceptable if it is corrected by growth factor or transfusion), and platelet count >= 100 x 10^9/L.
9. Adequate liver function as evidenced by bilirubin <= 1.5 times the upper limits of normal (ULN) and alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) <= 3 x ULN (in the case of liver metastases <= 5 x ULN), unless there are bone metastases, in which case liver specific alkaline phosphatase must be separated from the total and used to assess the liver function instead of the total alkaline phosphatase. In case alkaline phosphatase is >3 x ULN (in absence of liver metastases) or > 5 x ULN (in presence of liver metastases) AND patient is known to have bone metastases, the liver specific alkaline phosphatase must be separated from the total and used to assess the liver function instead of the total alkaline phosphatase.
10. Patients willing and able to comply with the study protocol for the duration of the study.
11. Written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.

EXCLUSION CRITERIA

1. Patients who have received any of the following treatments within the specified period before E7389 or TPC treatment start:

   * chemotherapy, radiation, trastuzumab or hormonal therapy within three weeks.
   * any investigational drug within four weeks.
2. Radiation therapy encompassing > 30% of marrow.
3. Prior treatment with mitomycin C or nitrosourea.
4. Pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen.
5. Patients with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study. Any signs (e.g., radiologic) and/or symptoms of brain metastases must be stable for at least 4 weeks before starting study treatment; radiographic stability should be determined by comparing a contrast-enhanced computed tomography or magnetic resonance imaging brain scan performed during screening to a prior scan performed at least 4 weeks earlier.
6. Patients with meningeal carcinomatosis.
7. Patients who are receiving anti-coagulant therapy with warfarin or related compounds, other than for line patency, and cannot be changed to heparin-based therapy if randomized to E7389 are not eligible. If a patient is to continue on mini-dose warfarin, then the prothrombin time (PT) or international normalized ratio (INR) must be closely monitored.
8. Women who are pregnant or breast-feeding; women of childbearing potential with either a positive pregnancy test at screening or no pregnancy test; women of childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception in the opinion of the Investigator. Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
9. Severe/uncontrolled intercurrent illness/infection.
10. Significant cardiovascular impairment (history of congestive heart failure > New York Heart Association grade II, unstable angina or myocardial infarction within the past six months, or serious cardiac arrhythmia).
11. Patients with organ allografts requiring immunosuppression.
12. Patients with known positive HIV status.
13. Patients who have had a prior malignancy, other than previous breast cancer, carcinoma in situ of the cervix, or non-melanoma skin cancer, unless the prior malignancy was diagnosed and definitively treated >= 5 years previously with no subsequent evidence of recurrence.
14. Patients with pre-existing neuropathy > Grade 2.
15. Patients with a hypersensitivity to halichondrin B and/or halichondrin B chemical derivative.
16. Patients who participated in a prior E7389 clinical trial whether or not E7389 was received.
17. Patients with other significant disease or disorders that, in the Investigator's opinion, would exclude the patient from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 762 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2009-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (137):
- United States (32):
  - US Oncology St. Vincent's Hospital - Bruno Cancer Center, Birmingham, Alabama
  - Bellflower Satellite, Bellflower, California
  - Research Center, Gilroy, California
  - US Oncology, Denver, Colorado
  - Florida Cancer Research Institute, Davie, Florida
  - Innovative Medical Research of South Florida, Inc., Miami, Florida
  - Peachtree Hematology/Oncology Consultants, PC, Atlanta, Georgia
  - US Oncology, Niles, Illinois
  - US Oncology, Indianapolis, Indiana
  - University of Iowa Hospital and Clinic, Iowa City, Iowa
  - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - Oncology Care Associates, P.L.L.C., Saint Joseph, Michigan
  - US Oncology, Columbia, Missouri
  - Montana Cancer Specialists, Missoula, Montana
  - US Oncology, Las Vegas, Nevada
  - US Oncology, Albany, New York
  - North Shore Hematology/Oncology Associates, East Setauket, New York
  - Weill Cornell Breast Cancer Center, New York, New York
  - Carolina Hematology Oncology Associates, Charlotte, North Carolina
  - US Oncology, Raleigh, North Carolina
  - US Oncology, Eugene, Oregon
  - St. Vincent Medical Center, Portland, Oregon
  - US Oncology, Bedford, Texas
  - US Oncology, Dallas, Texas
  - US Oncology, Houston, Texas
  - US Oncology, McAllen, Texas
  - US Oncology, Midland, Texas
  - US Oncology, Tyler, Texas
  - US Oncology, Spokane, Washington
  - Northwest Medical Specialists, Tacoma, Washington
  - US Oncology, Vancouver, Washington
  - US Oncology, Yakima, Washington
- Argentina (13):
  - Instituto Oncologico "Las Heras", Bahía Blanca, Buenos Aires
  - Hospital Britanico, C.a.b.a, Buenos Aires
  - Instituto FIDES especialidades Medicas, La Plata, Buenos Aires
  - Breast Clinica de la Mama, La Plata, Buenos Aires
  - CITEM, Quilmes, Buenos Aires
  - CER Instituto Medico, Quilmes Oeste, Buenos Aires
  - Instituto CAICI, Rosario, Pcia. Santa Fe
  - Centro Medico San Roque, San Miguel de Tucumán, San Miguel de Tucuman
  - Hosptial Interzonal General de Mar del Plata, Buenos Aires
  - Clinica Universitaria Privada Reina Fabiola, Córdoba
  - Sanatorio Frances, Córdoba
  - Instituto de Oncologia y Especialidades Medicas, Rosario Santa Fe
  - Clinica Especializada ISIS, Santa Fe
- Australia (6):
  - The Queen Elizabeth Hospital, Southport, Queensland
  - Servicio De Oncologia, Woodville South, South Australia
  - Maroondah Breast Clinic, Melbourne
  - Mater Medical Centre, North Sydney
  - Mount Hospital, Perth
  - Royal Perth Hospital, Department of Medical Oncology, Perth
- Austria (2):
  - Medizinische Universitatsklinik Graz, Graz Steiermark
  - Salzburger Landeskliniken Universitatsklinik fur Innere medizin III, Salzburg
- Belgium (5):
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Centre Hospitalier Notre-Dame - Reine Fabiola, Charleroi
  - UZ Gent, Ghent
  - AZ Groeninge, Campus Maria's Voorzienigheid, Kortrijk
- Brazil (9):
  - Centro Regional Integrado de Oncologia-CRIO, Fortaleza, Ceará
  - Centro de Pesquisas e Estudios do Centro Goiano, Giana, Goiás
  - Hospital Erasto Gaertner, Curitiba, Pará
  - Instituto Nacional do Cancer-Unidade III (INCA III), Rio de Janiero, Rio de Janeiro
  - CPO-Centro de Pesquisas em Oncologia, Porto Alegre, Rio Grande do Sul
  - CEPHO-Centro de Estudos e Pesquisa de Hematologia e oncologia, Santo André, São Paulo
  - Santo Andre Diagnosticos e Tratamentos, Santo André, São Paulo
  - Clinica de Oncologia Medica, São Paulo, São Paulo
  - Hospital Amaral Carvalho, Vila Assis, São Paulo
- Canada (3):
  - The Ottawa Hospital Regional Cancer Center, Ottawa, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - McGill University Health Centre, Department of Oncology, Gerald Bronfman Center, Montreal, Quebec
- Croatia (3):
  - Clinical Hospital Osijek, Osijek
  - University Hospital Center Zagreb, Zagreb
  - University Hospital for Tumors Zagreb, Zagreb
- Czechia (6):
  - Masaryk Memorial Cancer Institute, Brno
  - Hospital Jihlava, Jihlava
  - Clinic of Radiotherapy and Oncology, Prague
  - General Faculty Hospital Prague, Prague
  - Fakultni Thomayerova Nemocnice, Prague
  - Ustav radia ni onkologie 1. LF UK a FNB, Prague
- France (10):
  - Centre Paul Papin, Agners Cedex 01
  - Hopital Jean Minjoz, Besançon
  - Polyclinique Boredaux Nord Aquitaine, Bordeaux
  - Centre Francois Baclesse Caen, Caen
  - Centre Jean Perrin - CRLC, Clermont-Ferrand
  - Centre Georges-Francois Lecierc, Dijon
  - Hopital Edourad Herriot, Lyon
  - Institut Curie, Paris
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - Hopital Bretonneau, Tours
- Hungary (4):
  - Semmelweis Medical University, III. Dep. of Internal Med., Budapest
  - Debrecen Medical University, Department of Oncology, Debrecen
  - University of Pecs, Pécs
  - Markusovszky Teaching Hospital, Dept. of Oncoradiology, Sec. Med. Oncology, Szombathely
- Italy (7):
  - Azienda Ospedaliera Careggi, Firenze (FI)
  - Ospedale San Martino, Genova
  - Ospedale "Vito Fazzi" - Lecce, Lecce (LE)
  - Istituto Scientifico San Raffaele, Milan
  - Ospedale San Filippo Neri, Roma
  - Istituto Clinico Humanitas, Rozzano
  - UO di Oncologia, Sora
- Poland (7):
  - Akademickie Centrum Kliniczne Szpital Akademii Medycznej w, Gdansk
  - Szpital Morski im PCK w Gdyni Gdynskie Centrum Onkologii, Gdynia
  - Centrum Onkologii Instytut M. Sklodowskiej Curie w Warszawie Oddzial Gilwice, Gilwice
  - Centrum Onkologii Instytut M Sklodowskiej Curie, Oddzial w Krakowie, Krakow
  - Szpital Kiniczny Przemienienia Panskiego Uniwersyteu Medycznego im Karola Marcinkowskiego w Poznaniu, Poznan
  - Zachodniopomorski e Centrum, Szczecin
  - Centrum Onkologii Instytut im M. Sklodowskiej Curie w Warszawie, Warsaw
- Russia (13):
  - Republic Clinical Oncology Dispensary, Izhervsk Udmurtia
  - Kazan State Medical University, Kazan'
  - Krasnodar Territory Clinical Oncology Center, Krasnodar
  - Burdenko Main Military Hospital, Moscow
  - Nizhniy Novgorod City Oncology Center, Nizhny Novgorod
  - City Clinical Hospital #1, Novosibirisk
  - Republican Oncology Center, Petrozavodsk
  - State Institution of Healthcare Stavropol Region clinical Oncology dispensary, Pyatigorsk
  - Pavlov Medical University, Saint Petersburg
  - St Petersburg City Oncology Center, Saint Petersburg
  - NN Petrov Research Institute of Oncology, Saint Petersburg
  - Tomsk Regional Oncology Dispensary, Tomsk
  - GUZ YO Regional Clinical Oncology Hospital, Yaroslavl
- South Africa (4):
  - Panorama Medical Centre, Panorama, Cape Town
  - Eastern Cape Oncology Centre, GVI, St Georges Hospital, Port Elizabeth, Eastern Cape
  - Sandton Oncology Centre, Johannesburg
  - Pretoria Academic Hospital, Pretoria
- Spain (8):
  - Hospital Vall d Hebron, Barcelona
  - Hospital Mutua de Terrassa, Barcelona
  - Hospital Universitario de Girona Dr. Josep Trueta, Girona
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Unversitatio de Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital General Virgen del Rocio, Seville
  - Hospital Clinico de Zaragoza, Zanagoza
- Switzerland (5):
  - Kantonsspital Aarau, Aarau
  - Inselspital Bern, Bern Bern
  - Kantonsspital Oncology Haematology, Sankt Gallen
  - Spital Thun-Simmental AG, Thun
  - Kantonsspital Winterhur, Winterhur

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241
- [Derived] Miyoshi Y, Yoshimura Y, Saito K, Muramoto K, Sugawara M, Alexis K, Nomoto K, Nakamura S, Saeki T, Watanabe J, Perez-Garcia JM, Cortes J. High absolute lymphocyte counts are associated with longer overall survival in patients with metastatic breast cancer treated with eribulin-but not with treatment of physician's choice-in the EMBRACE study. Breast Cancer. 2020 Jul;27(4):706-715. doi: 10.1007/s12282-020-01067-2. Epub 2020 Mar 5. PMID 32133606
- [Derived] Wedam SB, Beaver JA, Amiri-Kordestani L, Bloomquist E, Tang S, Goldberg KB, Sridhara R, Ibrahim A, Kim G, Kluetz P, McKee A, Pazdur R. US Food and Drug Administration Pooled Analysis to Assess the Impact of Bone-Only Metastatic Breast Cancer on Clinical Trial Outcomes and Radiographic Assessments. J Clin Oncol. 2018 Apr 20;36(12):1225-1231. doi: 10.1200/JCO.2017.74.6917. Epub 2018 Mar 9. PMID 29522361
- [Derived] Twelves C, Cortes J, Kaufman PA, Yelle L, Awada A, Binder TA, Olivo M, Song J, O'Shaughnessy JA, Jove M, Perez EA. "New" metastases are associated with a poorer prognosis than growth of pre-existing metastases in patients with metastatic breast cancer treated with chemotherapy. Breast Cancer Res. 2015 Dec 9;17(1):150. doi: 10.1186/s13058-015-0657-1. PMID 27391598
- [Derived] Muss H, Cortes J, Vahdat LT, Cardoso F, Twelves C, Wanders J, Dutcus CE, Yang J, Seegobin S, O'Shaughnessy J. Eribulin monotherapy in patients aged 70 years and older with metastatic breast cancer. Oncologist. 2014 Apr;19(4):318-27. doi: 10.1634/theoncologist.2013-0282. Epub 2014 Mar 28. PMID 24682463
- [Derived] Cortes J, O'Shaughnessy J, Loesch D, Blum JL, Vahdat LT, Petrakova K, Chollet P, Manikas A, Dieras V, Delozier T, Vladimirov V, Cardoso F, Koh H, Bougnoux P, Dutcus CE, Seegobin S, Mir D, Meneses N, Wanders J, Twelves C; EMBRACE (Eisai Metastatic Breast Cancer Study Assessing Physician's Choice Versus E7389) investigators. Eribulin monotherapy versus treatment of physician's choice in patients with metastatic breast cancer (EMBRACE): a phase 3 open-label randomised study. Lancet. 2011 Mar 12;377(9769):914-23. doi: 10.1016/S0140-6736(11)60070-6. Epub 2011 Mar 2. PMID 21376385
- [Derived] Twelves C, Cortes J, Vahdat LT, Wanders J, Akerele C, Kaufman PA. Phase III trials of eribulin mesylate (E7389) in extensively pretreated patients with locally recurrent or metastatic breast cancer. Clin Breast Cancer. 2010 Apr;10(2):160-3. doi: 10.3816/CBC.2010.n.023. PMID 20299316

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 135 centers in 19 countries during the period of Nov 2006 to May 2009.
Groups:
- Eribulin Mesylate 1.4 mg/kg^2: Eribulin Mesylate 1.4 mg/kg^2 on Days 1 and 8
- Treatment of Physician's Choice: Treatment of Physician's Choice
Period: Overall Study
Arm/Group | Eribulin Mesylate 1.4 mg/kg^2 | Treatment of Physician's Choice
Started | 508 | 254
Completed | 24 | 10
Not Completed | 484 | 244
Not completed — Adverse Event | 50 | 24
Not completed — Progressive Disease | 336 | 153
Not completed — Clinical Progression | 61 | 36
Not completed — Withdrawal by Subject | 10 | 7
Not completed — Administrative | 6 | 9
Not completed — Physician Decision | 18 | 13
Not completed — Death | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eribulin Mesylate 1.4 mg/kg^2 | Treatment of Physician's Choice | Total
Number analyzed (Participants) | 508 | 254 | 762
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (10.34) | 55.9 (10.43) | 55.2 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 508 | 254 | 762
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 14 | 34
  White | 470 | 233 | 703
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Defined as the time from the date of randomization until the date of death from any cause.
Time Frame: From date of randomization until death from any cause
Population: Intent to Treat
Measure: Median (Full Range); unit: Days
Arm/Group | Eribulin Mesylate 1.4 mg/kg^2 | Treatment of Physician's Choice
Number analyzed (Participants) | 508 | 254
Days | 399 [360 to 434] | 324 [282 to 380]

2. Secondary Outcome: Progression-Free Survival.
Description: Measured using Response Evaluation Criteria in Solid Tumors (RECIST) and defined as the time from the date of randomization until progressive disease or death from any cause in the absence of of progressive disease.
Time Frame: Until disease progression or death.
Population: Intent to Treat
Measure: Median (Full Range); unit: Days
Arm/Group | Eribulin Mesylate 1.4 mg/kg^2 | Treatment of Physician's Choice
Number analyzed (Participants) | 508 | 254
Days | 113 [101 to 118] | 68 [63 to 103]

3. Secondary Outcome: Best Overall Response
Description: Measured by RECIST criteria and defined as the best response from the start of treatment until disease progression or recurrence. Lesions measured by computed tomography (CT) scan and magnetic resonance imaging (MRI). Objective response rate: complete response (CR-disappearance of all lesions)+ partial response (PR-30% decrease in lesion diameter), Progressive Disease (PD-20% increase in lesion diameter), stable disease (SD-neither shrinkage nor increase of lesions).
Time Frame: Until Day 30 or every 3 months during Follow-up period for patients who complete study without PD.
Population: Response Evaluable Population
Measure: Number; unit: Percent of Participants
Arm/Group | Eribulin Mesylate 1.4 mg/kg^2 | Treatment of Physician's Choice
Number analyzed (Participants) | 468 | 214
Percent of Participants
  Objective Response Rate (CR+PR) | 12.2 | 4.7
  Complete Response | 0.6 | 0
  Partial Response | 11.5 | 4.7
  Stable Disease | 44.4 | 44.9
  Progressive Disease | 40.6 | 49.1
  Not Evaluable | 2.6 | 1.4
  Unknown | 0.2 | 0

4. Secondary Outcome: Duration of Response.
Description: As measured by RECIST criteria and defined as the time from the first documented CR or PR until disease progression or death from any cause.
Time Frame: From first documented CR or PR until disease progression or death.
Population: Response Evaluable Population
Measure: Median (Full Range); unit: Days
Arm/Group | Eribulin Mesylate 1.4 mg/kg^2 | Treatment of Physician's Choice
Number analyzed (Participants) | 468 | 214
Days | 128 [116 to 152] | 205 [205 to 212]

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From start of study drug administration up to 30 days after the last dose of study drug (approximately up to 42 months)
Population: The safety analysis set was all participants who were randomized and who received at least a partial dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Eribulin Mesylate 1.4 mg/kg^2 | Treatment of Physician's Choice
Number analyzed (Participants) | 503 | 247
participants
  TEAE | 497 | 230
  SAE | 130 | 64

ADVERSE EVENTS:
Description: The safety analysis set was all participants who were randomized and who received at least a partial dose of study treatment.
Arm/Group | Eribulin Mesylate 1.4 mg/kg^2 | Treatment of Physician's Choice
Serious Adverse Events (participants affected / at risk) | 130/503 | 64/247
Other Adverse Events (participants affected / at risk) | 497/503 | 230/247
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate 1.4 mg/kg^2 (N=503) | Treatment of Physician's Choice (N=247)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Artery Thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 21 | 3
Neutropenia (Blood and lymphatic system disorders) | 9 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Asthenia/Fatigue (General disorders) | 7 | 6
Asthenia (General disorders) | 6 | 5
Pyrexia (General disorders) | 7 | 2
General Physical Health Deterioration (General disorders) | 6 | 2
Pain (General disorders) | 1 | 2
Performance Status Decreased (General disorders) | 0 | 3
Fatigue (General disorders) | 1 | 1
Mucosal Inflammation (General disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 2
Vomiting (Gastrointestinal disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Abdominal Pain (Gastrointestinal disorders) | 1 | 3
Ascites (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Colonic Obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Mouth Haemorrhage (Gastrointestinal disorders) | 1 | 0
Esophageal Stenosis (Gastrointestinal disorders) | 1 | 0
Esophageal Varices Haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Peritoneal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 1
Erysipelas (Infections and infestations) | 2 | 1
Catheter Related Infection (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 1
Lung Infection (Infections and infestations) | 2 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0
Aspergillosis (Infections and infestations) | 0 | 1
Breast Cellulitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Catheter Site Infection (Infections and infestations) | 1 | 0
Central Line Infection (Infections and infestations) | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Neutropenic Sepsis (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Staphylococcal Sepsis (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 7 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia/Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral Neuropathy (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 2 | 0
Lethargy (Nervous system disorders) | 2 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 1 | 0
Epiduritis (Nervous system disorders) | 1 | 0
Memory Impairment (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 1 | 0
Vocal Cord Paralysis (Nervous system disorders) | 0 | 1
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Metastases to Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Brain Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 3 | 2
Cardiovascular Insufficiency (Vascular disorders) | 1 | 1
Embolism (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Venous Thrombosis (Vascular disorders) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 1
Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Confusional State (Psychiatric disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 2
Hematuria (Renal and urinary disorders) | 0 | 1
Obstructive Uropathy (Renal and urinary disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 2 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 1
Bile Duct Obstruction (Hepatobiliary disorders) | 1 | 0
Cytolytic Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Body Temperature Increased (Investigations) | 2 | 1
Blood Creatinine Increased (Investigations) | 1 | 0
Palmar-Plantar Erythrodysaethesia Syndrome (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Ovarian Mass (Reproductive system and breast disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate 1.4 mg/kg^2 (N=503) | Treatment of Physician's Choice (N=247)
Asthenia/Fatigue (General disorders) | 273 | 99
Asthenia (General disorders) | 138 | 59
Fatigue (General disorders) | 148 | 47
Pyrexia (General disorders) | 107 | 31
Mucosal Inflammation (General disorders) | 44 | 25
Peripheral Edema (General disorders) | 46 | 21
Pain (General disorders) | 24 | 16
Nausea (Gastrointestinal disorders) | 175 | 70
Constipation (Gastrointestinal disorders) | 124 | 51
Diarrhea (Gastrointestinal disorders) | 96 | 45
Vomiting (Gastrointestinal disorders) | 94 | 44
Abdominal Pain Upper (Gastrointestinal disorders) | 46 | 15
Abdominal Pain (Gastrointestinal disorders) | 39 | 20
Dyspepsia (Gastrointestinal disorders) | 42 | 8
Stomatitis (Gastrointestinal disorders) | 38 | 12
Dry Mouth (Gastrointestinal disorders) | 29 | 3
Neutropenia (Blood and lymphatic system disorders) | 264 | 74
Anemia (Blood and lymphatic system disorders) | 97 | 56
Leukopenia (Blood and lymphatic system disorders) | 118 | 28
Peripheral Neuropathy (Nervous system disorders) | 174 | 40
Headache (Nervous system disorders) | 98 | 29
Paresthesia (Nervous system disorders) | 56 | 16
Peripheral Sensory Neuropathy (Nervous system disorders) | 62 | 10
Dizziness (Nervous system disorders) | 38 | 14
Neuropathy Peripheral (Nervous system disorders) | 39 | 9
Dysgeusia (Nervous system disorders) | 40 | 5
Arthralgia/Myalgia (Musculoskeletal and connective tissue disorders) | 112 | 29
Back Pain (Musculoskeletal and connective tissue disorders) | 81 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 73 | 13
Bone Pain (Musculoskeletal and connective tissue disorders) | 61 | 23
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 58 | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 54 | 17
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 37 | 15
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 38 | 11
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 38 | 10
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 27 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 225 | 24
Rash (Skin and subcutaneous tissue disorders) | 32 | 15
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 7 | 34
Urinary Tract Infection (Infections and infestations) | 49 | 13
Upper Respiratory Tract Infection (Infections and infestations) | 27 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 79 | 31
Cough (Respiratory, thoracic and mediastinal disorders) | 74 | 21
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 36 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 13
Weight Decreased (Investigations) | 107 | 36
Alanine Aminotransferase Increased (Investigations) | 27 | 6
Anorexia (Metabolism and nutrition disorders) | 101 | 32
Hypokalemia (Metabolism and nutrition disorders) | 36 | 5
Insomnia (Psychiatric disorders) | 38 | 10
Anxiety (Psychiatric disorders) | 27 | 11
Depression (Psychiatric disorders) | 27 | 3
Lacrimation Decreased (Eye disorders) | 35 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No